CLINICAL TRIAL: NCT05526677
Title: Effectiveness Evaluation of the Digital Workflow for Single-implant Immediate Loading
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-F(II)-20220117
Record Dates: First submitted 2022-08-04; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Single Missing Tooth Rehabilitation
Keywords: Single missing tooth; one-visit single-implant immediate loading; digital workflow; dynamic navigation; static surgical guide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dynamic navigation group or static guide group: Every patient has 2 missing in one jaw The missing tooth will be restored with one-visit single implant immediate loading.
  One implant placed is assisted with dynamic navigation system, and the other one is assisted with static surgical guide.
  Interventions: Device: x-guide dynamic navigation system

INTERVENTIONS:
Device: x-guide dynamic navigation system — One implant placement is assisted with x-guide dynamic navigation system. The other implant placement is assisted with static surgical guide
  Other Names: static surgical guide

SUMMARY:
Immediately implantation and immediate prosthesis could preserve the alveolar contour and gingival shape. The visiting time is quiet long. Pre-made prosthesis is a way to shorten the visiting time. But the implant has to be placed precisely. Novel digital workflow integrating dynamic navigation or static surgical guide to process one-visit single -implant immediate loading is possible. The study is to compare the x-guide dynamic navigation system or static guide system which one could assist the surgery more accuracy and place the prosthesis more smoothly.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 80 years old
* Miss two functional opposing teeth in one quadrant or the same jaw
* The situation of oral tissue satisfies the condition of implant immediate loading.

Exclusion Criteria:

* catastrophic illness,
* diabetes,
* cardiovascular diseases,
* osteoporosis,
* head and neck cancer,
* disabled
* pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient older than 18 years old, including both sexes. Every patient has 2 missing teeth in a jaw and one on each side. All the edentulous ridges suit the immediate loading criteria
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Record visiting time | during procedure
  Record the time (minutes) in every clinical procedure
Implant success rate | Change in periapical film of the implant on post operation immediately, post operation 1 month, 3 months, 6 months, 1 year
  No osteointegration of implant
Prosthesis success rate | Change in photo on post operation immediately, post operation 1 month, 3 months, 6 months, 1 year
  Morphology of the restoration
surgical complications | Post operation 1 week
  pain, swelling, infection after surgery
prosthetic success rates | Change in post operation immediately, post operation 1 month, 3 months, 6 months, 1 year
  final pink aesthetic score
Implant stability quotient (ISQ) | Change in post operation immediately, post operation 1 month, 3 months, 6 months, 1 year
  implant stability

SECONDARY OUTCOMES:
Type of incision | during the operation
  flap or flapless

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pozzi A, Arcuri L, Carosi P, Nardi A, Kan J. Clinical and radiological outcomes of novel digital workflow and dynamic navigation for single-implant immediate loading in aesthetic zone: 1-year prospective case series. Clin Oral Implants Res. 2021 Dec;32(12):1397-1410. doi: 10.1111/clr.13839. Epub 2021 Sep 8. PMID 34467555
- [Background] Lopes A, de Araujo Nobre M, Santos D. The Workflow of a New Dynamic Navigation System for the Insertion of Dental Implants in the Rehabilitation of Edentulous Jaws: Report of Two Cases. J Clin Med. 2020 Feb 4;9(2):421. doi: 10.3390/jcm9020421. PMID 32033089
- [Background] Block MS, Emery RW, Lank K, Ryan J. Implant Placement Accuracy Using Dynamic Navigation. Int J Oral Maxillofac Implants. 2017 Jan/Feb;32(1):92-99. doi: 10.11607/jomi.5004. Epub 2016 Sep 19. PMID 27643585
- [Background] Emery RW, Merritt SA, Lank K, Gibbs JD. Accuracy of Dynamic Navigation for Dental Implant Placement-Model-Based Evaluation. J Oral Implantol. 2016 Oct;42(5):399-405. doi: 10.1563/aaid-joi-D-16-00025. Epub 2016 Jun 6. PMID 27267658
- [Background] Dure M, Berlinghoff F, Kollmuss M, Hickel R, Huth KC. First comparison of a new dynamic navigation system and surgical guides for implantology: an in vitro study. Int J Comput Dent. 2021 Feb 26;24(1):9-17. PMID 34006059
- [Background] Block MS, Emery RW. Static or Dynamic Navigation for Implant Placement-Choosing the Method of Guidance. J Oral Maxillofac Surg. 2016 Feb;74(2):269-77. doi: 10.1016/j.joms.2015.09.022. Epub 2015 Sep 30. PMID 26452429